CLINICAL TRIAL: NCT04465539
Title: The Potential Therapeutic Role of Hydroxyethyl Starch and Hydrocortisone in Acute Aluminum Phosphide Poisoning: A Randamized Controlled Clinical Trial
Brief Title: The Potential Therapeutic Role of Hydroxyethyl Starch and Hydrocortisone in Acute Aluminum Phosphide Poisoning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HES & hydrocortisone
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Potential Therapeutic Role
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): received the standard ALP treatment according to TUPTC protocol as follows: patient resuscitation, care of airway, breathing and circulation, gastric decontamination with 2 ampoules sodium bicarbonate (each ampoule 25 ml containing 2.1 gm sodium bicarbonate) followed by activated charcoal in dose of 1 g/Kg orally, adequate hydration, normal saline administration (0.9% Sodium Chloride IV), vasopressors IV infusions, inhalation of 100% oxygen, ranitidine IV, magnesium sulfate IV infusion and other supportive treatment.
  Interventions: Drug: Placebo
- Hydroxyethyl starch group): (Experimental): Patients will start therapy with Hydroxyethyl starch instead of normal saline (6% hetastarch 600/0.75 in 0.9% sodium chloride) with a dose of 500 cc in 6 hours. Additionally, patient will receive the standard ALP treatment according to TUPTC protocol in the same order of placebo.
  Interventions: Drug: Hydroxyethyl Starch 130-0.4 60 MG/ML [Voluven]; Drug: Placebo
- Combined Hydroxyethyl starch and hydrocortisone group (Experimental): Patients will start therapy with combined Hydroxyethyl starch (Voluven®, fresenius kabi, Germany) and hydrocortisone (SOLU-CORTEF 100 mg ampoule) instead of normal saline of normal saline as follow: Hydroxyethyl starch dose is 6% hetastarch 600/0.75 in 0.9% sodium chloride with a dose of 500 cc in 6 hours. Hydrocortisone dose is 200-300 mg /day intravenously until normalization of blood pressure. Additionally, patient will receive the standard ALP treatment according to TUPTC protocol in the same order of placebo.
  Interventions: Drug: Hydroxyethyl Starch 130-0.4 60 MG/ML [Voluven]; Drug: Hydrocortisone; Drug: Placebo

INTERVENTIONS:
Drug: Hydroxyethyl Starch 130-0.4 60 MG/ML [Voluven] — Hydroxyethyl starch dose is 500 cc in 6 hours
  Arms: Combined Hydroxyethyl starch and hydrocortisone group; Hydroxyethyl starch group):
Drug: Hydrocortisone — Hydrocortisone dose is 200-300 mg /day intravenously
  Arms: Combined Hydroxyethyl starch and hydrocortisone group
Drug: Placebo — received the standard ALP treatment according to TUPTC protocol as follows: patient resuscitation, care of airway, breathing and circulation, gastric decontamination with 2 ampoules sodium bicarbonate (each ampoule 25 ml containing 2.1 gm sodium bicarbonate) followed by activated charcoal in dose of 1 g/Kg orally, adequate hydration, normal saline administration (0.9% Sodium Chloride IV), vasopressors IV infusions, inhalation of 100% oxygen, ranitidine IV, magnesium sulfate IV infusion and other supportive treatment.

SUMMARY:
Aluminum phosphide (ALP) is a widely used fumigant due to its efficiency as pesticides. It is available as tablets of Celphos, Alphos or Quickphos which are known as rice tablets. Each tablet weights 3 grams and contains 56% ALP and 44% of aluminum carbonate and paraffin. The incidence of ALP poisoning increased steadily specially in developing countries . ALP poisoning is considered to be one of the major causes of suicidal poisoning owing to its wide accessibility and low cost. However, accidental poisoning may occur during occupational exposure

DETAILED DESCRIPTION:
Aluminum phosphide (ALP) is a widely used fumigant due to its efficiency as pesticides. It is available as tablets of Celphos, Alphos or Quickphos which are known as rice tablets. Each tablet weights 3 grams and contains 56% ALP and 44% of aluminum carbonate and paraffin. The incidence of ALP poisoning increased steadily specially in developing countries . ALP poisoning is considered to be one of the major causes of suicidal poisoning owing to its wide accessibility and low cost. However, accidental poisoning may occur during occupational exposure.

Signs and symptoms of acute AlP poisoning include gastrointestinal, cardiovascular, hepatic, renal, and neurologic (1). Ingestion of ALP causes mild gastrointestinal (GIT) manifestations as nausea, vomiting, abdominal pain, in addition to chest tightness, hypotension, headache and dizziness. In severe cases, GIT hemorrhage, shock, severe metabolic acidosis, cardiac arrhythmia, convulsions and coma may occur. Later, signs of hepatic damage and renal insufficiency may develop.

Death usually occurs in 30-70% of cases within the first 24 hours resulting from refractory cardiogenic shock, cardiac arrhythmia, severe hypotension and metabolic acidosis.The main causes of cardiovascular collapse are increase capillary permeability, insufficient systemic vasoconstriction with low ventricular ejection fraction. On autopsy examinations, point to extravasation of fluid into the third space.

The management is exclusively supportive as gastric lavage with KMnO4 solution, treatment of hypotension and acidosis in view of the fact that there is no specific antidote available.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe acute aluminum phosphide poisoning
* systolic blood pressure (SBP) ≤90 mmHg
* PH ≤ 7.2
* HCO3 ≤15 meq/L
* during the first six hours of admission

Exclusion Criteria:

* Pregnant and lactating women
* Asymptomatic patients with history of acute aluminum phosphide exposure.
* Patients with co-ingestion to other substances in addition to aluminum phosphide.
* Patients with other major medical conditions (e.g. cardiovascular disease, renal or hepatic failure).
* Patients with previous medical intervention (fluid therapy and vasopressors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
mortality | 28 days from start of management
  mortality rate of patients

SECONDARY OUTCOMES:
Need for mechanical ventilation | Through study completion up to 6 months
  incidence of need for intubation and mechanical ventilation for each patient
need for ICU admission | Through study completion up to 6 months
  the incidence of need for ICU admission for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Abdel Hay, Tanta, El Gharbyia, Egypt